CLINICAL TRIAL: NCT00397462
Title: Blood Flow and Bone Density in Healthy Adult Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Binghamton University (Other)
Collaborators: Juvent, Inc (Industry); New york State Office of Science Technology and Academic Research (Unknown)
Responsible Party: Principal Investigator, Kenneth McLeod, Professor, BioEngineering, Binghamton University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSERC-005
Record Dates: First submitted 2006-11-07; First posted 2006-11-09 (Estimated); Results first posted 2016-09-26 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Bone Loss; Hypotensive; Lower Limb Fluid Pooling
Keywords: Osteoporosis; Sarcopenia; Calf muscle pump; Venous insufficiency; DEXA; Soleus muscle; APG
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis; Sarcopenia; Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): No change to usual behavior
- Low dose (Experimental): Request that calf muscle pump stimulation be used less than four hours per day
  Interventions: Device: calf muscle pump stimulation
- High dose (Experimental): Request that calf muscle pump stimulation be used at least four hours per day
  Interventions: Device: calf muscle pump stimulation

INTERVENTIONS:
Device: calf muscle pump stimulation — Micromechanical stimulation of the postural reflex arc to activate the soleus muscle to enhance lower limb fluid return to the heart
  Arms: High dose; Low dose

SUMMARY:
This project will test the efficacy of using a non-invasive neuromuscular stimulation on the plantar surface of the feet to prevent and/ or reverse bone loss in a sample of healthy adult women.

DETAILED DESCRIPTION:
Women between the ages of 30 and 60 years of age who work in positions that require them to be seated at desks for a large portion of each day, are capable of following the protocol for one year, have a t-score >- 2.5 (do not have osteoporosis), and respond to plantar stimulation will be asked to participate. Women will be excluded who are receiving medications for osteoporosis, taking hormone replacement therapy, taking steroids (either oral or inhaled), have metal implants in the tibia, hip and spine that interfere with DEXA (bone density) scanning, are professional or semi-professional athletes, have hyperparathyroidism, have a history of pulmonary embolism, deep vein thrombosis, peripheral vascular disease or varicose veins, have a Body Mass Index greater than 40 Kg/m2, have any type of neuromuscular disease, or are pregnant . Once the inclusion and exclusion criteria are met, 45 subjects will be randomized into 3 groups including 1) a group of 15 subjects who will use the device (stimulation) for up to 4 hours a day, 2) a group of 15 subjects that will use the device for up to 8 hours a day, and 3) a control group who will not use the device. Subjects in the two treatment groups will be asked to place their feet on a mechanical device that will deliver a slight vibration while they are seated at work. Vibrations between 30-60 Hz has been shown to stimulate the Meissner's corpuscles which in turn stimulate contraction of the deep muscles of the calves. This contraction has been shown to increase venous and lymphatic return from the lower extremities thus improve bone metabolism. Bone density readings and venous circulation will be measured at the onset of this research and will be repeated after 12 months of using the device.

ELIGIBILITY:
Inclusion Criteria:

* healthy women 30 - 60 years old
* work in seated positions

Exclusion Criteria:

* weigh more than 350 pounds
* pregnant or plan to become pregnant
* professional athlete
* currently on Hormone Replacement Therapy
* currently taking medication for osteoporosis
* currently on corticosteroids
* metal implants in tibia hip spine forearm
* diagnosed with hyperparathyroidism
* diagnosed with neuromuscular disease
* pulmonary embolism
* deep vein thrombosis
* peripheral vascular disease
* medications for hypertension

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2006-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth McLeod, PhD, Principal Investigator — Binghamton University SUNY, BioEngineering

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 Low Use: requested that they use the intervention during only the morning or afternoon up to 4 hours
- Group 2 High Use: requested that they use the intervention as much as possible during the work day
- Control: No intervention
Period: Overall Study
Arm/Group | Group 1 Low Use | Group 2 High Use | Control
Started | 16 | 13 | 15
Completed | 16 | 13 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: No use of the intervention
- Total: Total of all reporting groups
Arm/Group | Group 1 Low Use | Group 2 High Use | Control | Total
Number analyzed (Participants) | 16 | 13 | 15 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 13 | 15 | 44
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (8.1) | 44.8 (9.1) | 44.5 (8.1) | 45.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 15 | 44
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 13 | 15 | 44

OUTCOME MEASURES:

1. Primary Outcome: Bone Density of Proximal Femur
Description: Proximal femur bone mineral density by dual energy x-ray absorptiometry (DXA)
Time Frame: One year
Measure: Mean (Standard Error); unit: percent change in bone density
Arm/Group | Control | Low Dose | High Dose
Number analyzed (Participants) | 15 | 16 | 13
percent change in bone density | -0.133 (.370) | -.675 (.437) | 1.3 (0.382)

2. Secondary Outcome: Proximal Tibia Bone Density
Description: Proximal tibia bone mineral density by dual energy x-ray absorptiometry (DXA)
Time Frame: One year
Measure: Mean (Standard Error); unit: percent change in bone density
Arm/Group | Control | Low Dose | High Dose
Number analyzed (Participants) | 15 | 16 | 13
percent change in bone density | 1.14 (1.14) | -2.111 (.64) | 1.65 (.56)

ADVERSE EVENTS:
Groups:
- Control: did not use the intervention
Arm/Group | Group 1 Low Use | Group 2 High Use | Control
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/13 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No